CLINICAL TRIAL: NCT07261995
Title: Comparison of Outcomes of Extracorporeal Shock Wave Lithotripsy Versus Retrograde Intrarenal Surgery in the Management of Renal Calculi Measuring 1 to 2 Centimeters
Brief Title: Comparison of Extracorporeal Shock Wave Lithotripsy Versus Retrograde Intrarenal Surgery in the Management of Renal Calculi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Waqas Arshad, Principal Investigator, Ziauddin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ziauddin Uro1
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Nephrolithiasis; Renal Calculi
Keywords: Kidney stones; Nephrolithiasis; Urolithiasis; Extracorporeal shock wave lithotripsy; Retrograde intrarenal surgery
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Urolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESWL (Active Comparator): Patients with a single renal stone measuring 1-2 centimeters receive extracorporeal shock wave lithotripsy (ESWL) as a day-care outpatient procedure under sedation. Shock waves are delivered starting at 60 impulses per minute and titrated up to 100 impulses per minute according to patient tolerance, with a maximum of 3000 shocks per session. Standard peri-procedural care, analgesia, hydration advice, and antibiotic prophylaxis according to institutional protocol are provided.
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL)
- Group RIRS (Active Comparator): Patients with a single renal stone measuring 1-2 centimeters undergo retrograde intrarenal surgery (RIRS) under general anesthesia. All patients are pre-stented with a 5 Fr double-J ureteral stent 2-3 weeks prior to the definitive procedure. A flexible ureteroscope is advanced to the renal collecting system through a ureteral access sheath, and the stone is fragmented using a Holmium:YAG laser with energy 0.5-1.2 Joules and frequency 20-40 Hertz (dusting or fragmentation technique as appropriate). A double-J stent is left in situ at the end of the procedure and scheduled for removal after three weeks. Standard postoperative care is provided.
  Interventions: Procedure: Retrograde Intrarenal Surgery (RIRS)

INTERVENTIONS:
Procedure: Extracorporeal Shock Wave Lithotripsy (ESWL) — Extracorporeal shock wave lithotripsy delivered as an outpatient procedure under sedation, using a standard lithotripter. Shock waves are applied at 60-100 impulses per minute, up to a maximum of 3000 shocks per session, to fragment a 1-2 centimeter renal calculus. Patients receive standard analgesia, hydration counselling, and antibiotic prophylaxis according to hospital protocol.
  Other Names: Shock wave lithotripsy
  Arms: Group ESWL
Procedure: Retrograde Intrarenal Surgery (RIRS) — Retrograde intrarenal surgery performed under general anesthesia after prior placement of a 5 Fr double-J ureteral stent. A flexible ureteroscope introduced via the urethra and ureteral access sheath is used to visualise the renal stone. Stone disintegration is achieved with a Holmium:YAG laser (0.5-1.2 Joules, 20-40 Hertz) using dusting or fragmentation, followed by placement of a double-J stent for three weeks. Standard postoperative analgesia, antibiotics, and hydration advice are given.
  Arms: Group RIRS

SUMMARY:
This study is being carried out in patients with kidney stones measuring between 1 and 2 centimeters. Kidney stones are common in Pakistan and can cause severe pain, infection, and repeated hospital visits. Two commonly used treatments for stones of this size are extracorporeal shock wave lithotripsy (ESWL) and retrograde intrarenal surgery (RIRS). ESWL uses shock waves applied from outside the body to break the stone into small fragments that can pass in the urine. RIRS is a minimally invasive endoscopic procedure in which a thin flexible scope is passed through the urinary passage into the kidney and a laser is used to break the stone.

Adult patients aged 18 to 65 years with a single kidney stone of 1-2 cm will be included. According to the urologist's clinical judgment and patient preference, individuals will undergo either ESWL (Group A) as a day-care shock wave procedure or RIRS (Group B) under general anesthesia using a laser. All patients will receive standard care before and after the procedure and will be followed for 28 days.

The study will compare how completely the stone is cleared (based on a CT scan), how long patients stay in hospital, how much pain they feel after the procedure, and whether they develop visible blood in the urine or signs of infection such as fever and raised white cell count. The need for any further procedure for the same stone will also be recorded. The central hypothesis is that there is a meaningful difference between ESWL and RIRS in stone clearance, safety, pain, and need for retreatment. The findings are expected to help doctors and patients choose the most suitable treatment for kidney stones of this size in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.
* Patients diagnosed with a single renal calculus measuring between 1 cm and 2 cm, confirmed on imaging (ultrasound or non-contrast CT KUB).

Exclusion Criteria:

* Presence of multiple renal stones or bilateral renal stones.
* Patients with anatomical abnormalities such as horseshoe kidney, ureteropelvic junction obstruction, or calyceal diverticulum based on medical history or radiological findings.
* Active urinary tract infection at the time of intervention.
* Pregnant women.
* Patients with bleeding disorders or on anticoagulation therapy that cannot be safely stopped.
* Patients with chronic kidney disease (eGFR < 30 mL/min/1.73 m²).
* Patients with morbid obesity (BMI > 40 kg/m²).
* Patients with solitary kidney.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Stone clearance rate | 28 days after the procedure
  Proportion of participants in each treatment group who achieve successful stone clearance, defined as absence of visible stone or presence of a clinically insignificant residual fragment measuring ≤4 mm on non-contrast computed tomography of kidneys, ureters and bladder (CT-KUB). All scans will be interpreted and reported by a consultant radiologist blinded to treatment allocation. Stone clearance will be analysed as a binary variable (cleared/not cleared) for comparison between extracorporeal shock wave lithotripsy and retrograde intrarenal surgery.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS score) | At 24 hours after the procedure
  Patient-reported pain severity measured on a 10-cm Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents worst imaginable pain. Scores will be recorded by trained nursing staff and compared between groups as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Waqas Arshad, Principal Investigator — Ziauddin Universty
Locations (1):
- Ziauddin Hospital, Karachi, Sindh, Pakistan